CLINICAL TRIAL: NCT01817179
Title: Effects of Functional Electrical Stimulation Neuroprosthesis in Children With Hemiplegic Cerebral Palsy
Brief Title: Functional Electrical Stimulation for Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN001-Effects of FES/PwP
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2013-03

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: hemiplegia, cerebral palsy, neuroprosthesis, children
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FES neuroprosthesis to dorsiflexors on affected side (Experimental): Participants will use FES neuroprosthesis to dorsiflexors on affected leg for 3 months at home.
  Interventions: Other: FES neuroprosthesis to dorsiflexors on affected leg

INTERVENTIONS:
Other: FES neuroprosthesis to dorsiflexors on affected leg
  Other Names: Bioness L300

SUMMARY:
The purpose of this study is to evaluate how a functional electrical stimulation (FES) device worn on the lower leg effects how children (ages 6-17 years) with hemiplegic cerebral palsy walk and perform other functional activities.

The investigators expect to find that wearing the functional electrical stimulation device will improve walking and other functional activities of children with hemiplegic cerebral palsy. Participants will be trained in use of the device and will be required to wear it daily for 3 months. Each participant will be evaluated before beginning the intervention and after completing the intervention. This study will provide important information regarding the benefits of this treatment intervention in children with hemiplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemiplegic Cerebral Palsy
* Gross Motor Function Classification System (GMFCS) I or II
* Age 6-17 years inclusive
* Demonstrate foot drop during gait without wearing ankle foot orthosis
* Tolerance to neuroprosthesis stimulation
* Physician referral to participate in intervention
* Passive dorsiflexion to at least neutral with knee extended
* Available to travel to and from study visits
* Ability to follow instructions and cooperate with study protocol
* Caregiver reads and understands English

  * Exclusion criteria:
* Any metal implants containing electrical circuitry
* Continuous regular use of neuroprosthesis stimulation previous to study enrollment
* Previous orthopaedic procedure involving tibialis anterior muscle at any time
* Previous orthopaedic procedure to affected limb in the last year
* Botulinum toxin administered within the past 3 months, or plans for such treatment during the course of the study
* Any condition that PI feels would limit ambulatory progress (e.g. arthritis, uncontrolled seizures)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
peak ankle dorsiflexion range during swing phase in gait | will be assessed at baseline and 3 months after continous use of neuroprosthesis

SECONDARY OUTCOMES:
gait efficiency | after 3 months of neuroprosthesis use

OTHER OUTCOMES:
functional skills | at baseline and 3 months after neuroprosthesis use
  will included timed up and downs stairs,six minute walk test, and an obstacle course

CONTACTS AND LOCATIONS:
Overall Officials: Amy F Bailes, PT, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States